CLINICAL TRIAL: NCT01490957
Title: Functional Assessment of Cancer Therapy - Bone Marrow Transplant (FACT-BMT)
Brief Title: Functional Assessment of Cancer Therapy - Bone Marrow Transplant
Acronym: FACT-BMT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: RAC# 2071-079; RAC# 2071-079
Record Dates: First submitted 2011-12-11; First posted 2011-12-13 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Hodgkin Disease; Lymphoma, Non-Hodgkin
Keywords: HD; NHL
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Database Management Systems; RTEL1 protein, human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Database — Database
  Other Names: Database of Newly Diagnosed HD and NHL

SUMMARY:
Functional Assessment of Cancer Therapy - Bone Marrow Transplant

DETAILED DESCRIPTION:
Functional Assessment of Cancer Therapy - Bone Marrow Transplant (FACT-BMT)

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed Hodgkin's Disease and Non-Hodgkin's Lymphoma

Exclusion Criteria:

* Patients with diagnosis other than HD and NHL.

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Lymphoma database
Sampling Method: Non-Probability Sample
Enrollment: 113 (Estimated)
Dates: Start 2008-03

CONTACTS AND LOCATIONS:
Overall Officials: A Al-Zahrani, M.D., Principal Investigator — KFSH & RC
Locations (1):
- Kfsh & Rc, Riyadh, Saudi Arabia